CLINICAL TRIAL: NCT06274567
Title: Targeting Emotion Regulation in Bipolar Disorder With Intermittent Theta Burst Stimulation: A Mechanistic Study
Brief Title: Intermittent Theta Burst Stimulation (iTBS) for Emotion Regulation in Bipolar Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Kristen K. Ellard, Ph.D., Assistant Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024P000348
Record Dates: First submitted 2024-02-13; First posted 2024-02-23 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Randomized allocation
Who Masked: Participant, Care Provider, Investigator
Masking Description: We will use an active/placebo TMS coil. TMS operator and participant will be blinded to active versus sham. Investigator will be blinded to participant condition assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active intermittent theta burst stimulation (iTBS) (Experimental): The Active intermittent theta burst stimulation (iTBS) arm will receive active iTBS applied to the inferior parietal lobule (IPL)
  Interventions: Device: Transcranial Magnetic Stimulation (TMS)
- Sham intermittent theta burst stimulation (iTBS) (Placebo Comparator): The Sham intermittent theta burst stimulation (iTBS) arm will receive sham iTBS applied to the inferior parietal lobule (IPL)
  Interventions: Device: Sham (placebo) TMS

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation (TMS) — Transcranial magnetic stimulation (TMS) is a non-invasive tool for modulating patterns of brain activation and circuit connectivity. It uses electromagnetic pulses to induce electric currents over the cortex that serve to depolarize or hyperpolarize neurons, thereby changing patterns of synaptic activity. This study uses intermittent theta burst stimulation (iTBS), an efficient TMS protocol that uses high frequency (50Hz) triplets of TMS given every 200 milliseconds (i.e. at 5 Hz).
  Arms: Active intermittent theta burst stimulation (iTBS)
Device: Sham (placebo) TMS — Sham stimulation works by blocking the magnetic field with an internal spacer on the sham side of the TMS coil, allowing the operator to place the coil surface against the scalp. A brief electric pulse calibrated to the stimulator output is delivered to the scalp simultaneous to the TMS pulse to mimic the scalp sensation during the sham condition. 75 Importantly, the electric pulse is calibrated to the stimulator output to ensure a realistic sham condition.
  Arms: Sham intermittent theta burst stimulation (iTBS)

SUMMARY:
The objective of this study protocol is to test whether intermittent theta-burst transcranial magnetic stimulation (iTBS-TMS) to the inferior parietal lobule (IPL) can strengthen functional connectivity with a key region in emotion regulation (ER) neurocircuitry (anterior insula, AI) and improve performance on ER-related tasks in patients with bipolar disorder. Individual IPL sites for stimulation will be identified through baseline, pre-TMS functional magnetic resonance imaging (fMRI) scans. Patient-specific IPL subregions showing positive functional connectivity with the anterior insula and falling within the patient-specific frontoparietal control network will be used as individualized target sites for TMS stimulation. Patients will be randomized to receive 24 sessions of active versus sham iTBS to patient-specific IPL targets (6 sessions/day, 4 days, 43,200 pulses total). Post-iTBS resting-state and task-based fMRI scans will be acquired 3 days after the final day of iTBS administration (Day 4) following identical procedures as baseline. Effects of iTBS-TMS on ER will be evaluated by comparing pre-TMS versus post-TMS functional connectivity and behavior during performance on ER tasks.

DETAILED DESCRIPTION:
The specific goal of this mechanistic study is to test whether targeted engagement of the inferior parietal lobule (IPL) using a rapid and robust form of transcranial magnetic stimulation, accelerated intermittent theta burst stimulation (aiTBS), will increase emotion regulation (ER) in patients with bipolar disorder (BD). Specifically, the Investigators will experimentally test whether stimulation the IPL with aiTBS can strengthen functional neurocircuitry supporting healthy ER, as indexed by increased IPL and anterior insula (AI) functional connectivity and improved performance on ER-related behavioral tasks. The Investigators will use computer tasks that measure ER and functional magnetic resonance imaging (fMRI) to examine changes in brain function and behavior following real versus sham aiTBS in individuals with BD. Patients will be randomized to either active or sham aiTBS and will receive 6 sessions of high dose (1800 pulses) iTBS per day over a course of 4 days (24 sessions total). Patients will be scanned at baseline and 3 days after Day 4 of aiTBS in order to examine ER-related neuroplastic effects of IPL stimulation. To increase the potential clinical utility of findings from this study, the Investigators will examine the effects of aiTBS to the IPL in a sample of BD patients who are currently depressed, the most common and chronic mood state in this population. Following informed consent, all participants will complete a battery of self-report questionnaires assessing ER and will complete a computer-based ER task (Balloon Analog Risk Task; BART). Participants will then complete a functional magnetic resonance imaging (fMRI) scanning session consisting of (1) structural, (2) resting state, and (3) task-based (Affective Multisource Interference Task; MSIT-IAPS) scans. Participants will then be randomized to either Active (n=60, 30 per site) or Sham (N=60, 30 per site) aiTBS conditions in a double-blind design. Both Active and Sham procedures will consist of 4 days of iTBS (6 sessions/day). Participants will repeat the BART computer-based task and fMRI scanning procedures (structural, resting state, MSIT-IAPS in scanner task) within 3 days after Day 4 stimulation to measure the neuroplastic effects of aiTBS. The Investigators propose to recruit 136 individuals with a diagnosis of BD and a current depressed episode. The study will have 68 per each of the two groups (Active, Sham) at baseline and anticipate approximately 10% loss to attrition by post aiTBS. As the study has a single primary outcome (aiTBS-induced changes in IPL-AI functional connectivity), the Investigators use an alpha-level (Type 1 error rate) of 0.05. In preliminary data (n=8), the Investigators observed an increase in IPL-AI functional connectivity from 0.04 (SD=0.17) to 0.15 (SD=0.22), with correlation of 0.80 after a single day of 10 sessions active iTBS, corresponding to an effect size of Cohen's d=0.57. The Investigators anticipate a small "placebo" effect in the TBS group, of about d=0.10, and conservatively assume a correlation of 0.65, rather than the 0.80 seen in the pilot study. With these assumptions, the study has 80% power for an active aiTBS effect of 0.45, relative to sham aiTBS. The Investigators note that these effect size estimates are based on a much smaller dose of iTBS than the dose to be administered in the proposed study (18,000 pulses versus 43,200 pulses) - thus, it is plausible that the effect sizes seen in the study will be larger than those in the pilot data. See "Statistical Design and Power" for full details of data analysis plan.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals of all genders
2. ages 24-65
3. Diagnostic Statistical Manual (DSM-5) defined diagnosis of bipolar I or II disorder (BD); assessed using the Mini-International Neuropsychiatric Interview (M.I.N.I.) version 7.0.2.
4. Current depressive episode, assessed using the Montgomery-Asberg Depression Rating Scale (MADRS) score ≥20,
5. Ability to provide informed consent and verifiable contact information, including current psychiatric treatment provider
6. Stable medication regimen for at least one month, which must include a mood stabilizer

Exclusion Criteria:

1. current mania/hypomania assessed by the Young Mania Rating Scale (YMRS > 12)
2. rapid-cycling bipolar illness, defined as >4 episodes per year, indicating increased risk of switch to mania
3. current active suicidality (suicidal ideation with intent or plan), as assessed by a score >4 on the MADRS item #10
4. current substance use disorder for the past 6 months; substance use disorder in remission permitted
5. history of psychosis
6. dementia or other major neurological disorders, as assessed by a Mini-Mental State Exam (MMSE) score <24 and Montreal Cognitive Assessment (MOCA) score <26
7. medical illness or non-psychiatric medical treatment that would likely interfere with study participation
8. contraindications for magnetic resonance imaging (MRI) or transcranial magnetic stimulation (TMS), including the presence of metallic implants that would interfere with safety (i.e. cardiac pacemaker, metal plates, non-removable body piercings, etc.), history of seizure disorder, history of head trauma
9. a clinical course of a neuromodulatory therapy (e.g. transcranial magnetic stimulation, transcranial direct current stimulation, electroconvulsive therapy) within the past 6 months
10. current use of benzodiazepines, which can interfere with iTBS stimulation
11. current pregnancy, to limit potential risks to an unborn child

Other: Given that >86% of BD patients experience lifetime comorbid anxiety, co-occurring anxiety disorders will be allowable for inclusion, thus providing a more representative sample of bipolar patients who typically present at our Clinics for treatment. Comorbid anxiety disorders are not a criteria for inclusion or exclusion.

Ages: 24 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2024-09-20 (Actual); Primary Completion 2029-02-28 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Correlated functional magnetic resonance imaging (fMRI) time series (functional connectivity) | Baseline, 1-3 days post 4-day intervention (up to 4 weeks post Baseline)
  Primary outcome will be changes in the correlated time series between brain regions (inferior parietal lobule and anterior insula) from baseline to post intervention

SECONDARY OUTCOMES:
Affective Multisource Interference Task | Baseline, 1-3 days post 4-day intervention (up to 4 weeks post Baseline)
  Secondary outcome will be changes in reaction time responses to an affective interference task
Balloon Analogue Risk Task | Baseline, 1-3 days post 4-day intervention (up to 4 weeks post Baseline)
  Secondary outcome will be changes in number of button presses in response to a risk versus reward task

CONTACTS AND LOCATIONS:
Overall Officials: Kristen K Ellard, PhD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Martinos Center for Biomedical Imaging, Charlestown, Massachusetts
  - University of Pennsylvania, Center for Neuromodulation in Depression and Stress, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No